CLINICAL TRIAL: NCT06815523
Title: Prediction of Duration of Mechanical Venylation in Patients Wit Acute Hypoxemic Respiratory Failure Usinf Machine Learning Approaches
Brief Title: Prediction of Duration of Mechanical Ventilation in Acute Hypoxemic Respiratoty Failure
Acronym: PREMIER
Status: Active, not recruiting | Type: Observational
Sponsor: Jesus Villar (Other)
Collaborators: Hospital Universitario Dr. Negrín (Las Palmas de Gran Canaria) (Unknown); Iinstituto de Salud Carlos III (Unknown)
Responsible Party: Sponsor-Investigator, Jesus Villar, Scientific Advisor, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: PIFIISC24
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: mechanical ventilation; machine learning; prediction of prolonged mechanical ventilation; outcome
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Machine Learning; Logistic Models

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation/testing cohort: The investigators will use a chort of 75% of patients, randomly selected, with data at T0, T24 and T48 after diagnosis of acute hypoxemic respiratory failure (AHRF). We will apply machine learning approaches.
  Interventions: Other: Machine learning and logistic regression for the training/testing cohort and validation cohort
- Validation hohort: we will use 25% of unseen patients, randomly selected, with data at T0, T24 and T48 after diagnosis of AHRF.
  Interventions: Other: Machine learning and logistic regression for the training/testing cohort and validation cohort

INTERVENTIONS:
Other: Machine learning and logistic regression for the training/testing cohort and validation cohort — Machine learning and logistic regression for the validation cohort

SUMMARY:
Acute hypoxemic respiratory failure (AHRF) is a common cause of admission in intensive care units (ICUs) worldwide. We will assess machine learning (ML) techniques for prediction of prolonged duration (> or = to 7 days) of mechanical ventilation (MV) in 1,241 patients enrolled in the PANDORA study in Spain. The study was registered with ClinalTrials.gov (NCT03145974). Our aim is to identify a model with the minimum number of variables that predict duration of prolonged ventilation in AHRF patients using data as early as from the first 48 hours with machine learning algorithms.

DETAILED DESCRIPTION:
Acute hypoxemic respiratory failure (AHRF) is the most common cause of admission in intensive care units (ICUs) worldwide. The investigators will assess the value of machine learning (ML) techniques for prediction of prolonged duration (> or equeal to 7 days) of mechanical ventilation (MV) in 1,241 patients enrolled in the PANDORA study in Spain. Few studies have investigated the prediction of prolonged MV in patients with AHRF.

For model training and testing, the investigators will extract data from random pateints from the first 2 days after diagnosis of AHRF. The investigators had a database with 2,000,000 anonymized and dissociated demographics and clinically relevant data from 1,241 patients with AHRF from 22 hospitals in Spain. The investigators will follow the TRIPOD guidelines for prediction models. The investigators will screen relevant collected variables using a genetic algorithm variable selection to achieve parsimony. We will use 5-fold corss-validation in the data set of patients with data at T0, T24 and T48. We will use 25% of patients randomly selected for evaluation of the model.

ELIGIBILITY:
Inclusion Criteria:

* enotracheal intubation puls mechanical ventilation
* PaO2/FiO2 ratio <or = 300 mmHg under MV with PEEP >or =5 and FiO2 >or = 0.3

Exclusion Criteria:

* Brain death patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: De-identified dataset inclusing 1241 ventilated patients with AHRF admitted in a network of Spainisg ICUs.
Sampling Method: Non-Probability Sample
Enrollment: 1241 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
MV duration | up to 100 weeks
  duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Villar, Study Director — Fundacion Canaria Instituto de Investigación Sanitaria de Canarias
Locations (2):
- Spain (2):
  - Hospital Dr. Negrin, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No
Ethical reasons

REFERENCES:
- [Derived] Villar J, Gonzalez-Martin JM, Fernandez C, Soler JA, Rey-Abalo M, Mora-Ordonez JM, Ortiz-Diaz-Miguel R, Fernandez L, Murcia I, Robaglia D, Anon JM, Ferrando C, Parrilla D, Dominguez-Berrot AM, Cobeta P, Martinez D, Amaro-Harpigny A, Andaluz-Ojeda D, Fernandez MM, Gomez-Bentolila E, Steyerberg EW, Camporota L, Szakmany T. Predicting Outcome and Duration of Mechanical Ventilation in Acute Hypoxemic Respiratory Failure: The PREMIER Study. J Clin Med. 2025 Nov 7;14(22):7903. doi: 10.3390/jcm14227903. PMID 41302939